CLINICAL TRIAL: NCT04038099
Title: Lessons on Urethral Lidocaine in Urodynamics (LULU): Impact of Intraurethral Lidocaine on Cystometric Parameters and Discomfort
Brief Title: Lessons on Urethral Lidocaine in Urodynamics
Acronym: LULU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christina Hegan, Nurse practitioner, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STU-2019-0540
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Urethra Issue; Pelvic Organ Prolapse; Urinary Incontinence; Vaginal Vault Prolapse; Cystocele; Uterine Prolapse; Vaginal Prolapse; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Cystocele; Uterine Prolapse; Pelvic Floor Disorders | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Water Based Lubricating Jelly (Placebo Comparator): 5ml of Water Based Lubricating Jelly
  Interventions: Drug: Water-Based Vaginal Lubricant
- Lidocaine 2% Jelly (Active Comparator): 5ml of Lidocaine 2% Jelly
  Interventions: Drug: lidocaine topical

INTERVENTIONS:
Drug: Water-Based Vaginal Lubricant — 5cc water based jelly applied intraurethral
  Arms: Water Based Lubricating Jelly
Drug: lidocaine topical — 5cc 2% lidocaine jelly applied intraurethral
  Arms: Lidocaine 2% Jelly

SUMMARY:
This trial will assess whether use of intraurethral 2% lidocaine jelly meaningfully impacts sensation during filling (i.e., a change of more than 25% of first sensation, first desire to void, strong desire to void, or maximum cystometric capacity) and determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts pain/discomfort, filling metrics, and voiding metrics.

DETAILED DESCRIPTION:
This trial is a randomized, double blind, controlled trial for patients undergoing complex cystometric evaluation. Patients will undergo routine complex cystometric evaluation for acquisition of baseline data using a small amount of intraurethral aqueous jelly for catheter lubrication. Then, they will be randomized to instillation of either placebo (additional intraurethral aqueous jelly, 5ml) or intraurethral 2% lidocaine jelly. Participants then undergo complex cystometry a second time. Normal variations in studies with placebo will be compared to variations within the 2% lidocaine jelly group to determine if cystometric parameters are altered in any clinically important ways. Patient discomfort will also be evaluated by both the patient and the urodynamics advanced practice nurse.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* >18 years of age
* Already scheduled (or being scheduled) for UDS to assess urinary incontinence
* Able to speak and read in English

Exclusion Criteria:

* Diagnosis of pelvic pain, interstitial cystitis, or bladder pain syndrome
* Known neurogenic disease impacting voiding/ continence (e.g., Parkinson disease, multiple sclerosis, myasthenia gravis, recent stroke)
* Active UTI
* Pelvic organ prolapse that is unable to be easily reduced
* Pregnancy or breastfeeding
* Allergy or hypersensitivity to lidocaine or local anesthetics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 63 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Hegan, APRN WHNP-BC, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Result] Hicks, C., Schaffer, J., Pruzynski, J., & Rahn, D. (2022). Impact of Intraurethral Lidocaine on Cystometric Parameters and Patient Discomfort: A Randomized Controlled Trial. Urologic Nursing, 42(5), 237-257. https://doi.org/10.7257/2168-4626.2022.42.5.237
- See also: Research Video — https://vimeo.com/792762166/20321831a7

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (11.2) | 60.2 (11.4) | 61.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 63
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 23 | 21 | 44
  Black, non-Hispanic | 4 | 5 | 9
  Hispanic | 2 | 5 | 7
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63
Insurance Type [Count of Participants; unit: Participants] — One participant in the water based lubricant group had both Medicare and private insurance.
  Participants
    Private | 16 | 21 | 37
    Medicare | 14 | 12 | 26
    Self-pay | 1 | 0 | 1
Current smoker [Count of Participants; unit: Participants] | 3 | 3 | 6
Parous [Count of Participants; unit: Participants] | 27 | 29 | 56
Prior surgery for Stress Urinary Incontinence (SUI) [Count of Participants; unit: Participants] | 5 | 7 | 12
Prior surgery for prolapse [Count of Participants; unit: Participants] | 3 | 4 | 7
Prior hysterectomy [Count of Participants; unit: Participants] | 14 | 14 | 28
>3 UTIs in the past year [Count of Participants; unit: Participants] | 4 | 2 | 6
Diabetes [Count of Participants; unit: Participants] | 2 | 4 | 6
Stage of most severely prolapsed compartment [Count of Participants; unit: Participants] — Stages of prolapse were graded using the pelvic organ prolapse staging system as follows:
  Stage 0 - No prolapse.
  * Stage I - the most distal portion of the prolapse is >1 cm proximal to the level of the hymenal plane
  * Stage II - The most distal portion of the prolapse is between ≤1 cm proximal to the hymenal plane and ≤1 cm distal to the hymenal plane
  * Stage III - The most distal portion of the prolapse is between >1 cm distal to the hymenal plane, but no further than 2 cm less than the total vaginal length in centimeters
  * Stage IV - Eversion of the total length of the vagina.
  Participants
    Stage 0 or 1 | 12 | 9 | 21
    Stage 2 | 12 | 9 | 21
    Stage 3 or 4 | 6 | 14 | 20
Detrusor overactivity on UDS #1 [Count of Participants; unit: Participants] — Presence or absence of bladder detrusor overactivity (bladder spasm) during urodynamic bladder test #1.
  Participants | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Sensation as Indicated by the Volume of Water Filled (ml) at the Time of Patient Perception of First Sensation, First Urge to Void, Strong Urge to Void, and Full Bladder Capacity During Bladder Filling.
Description: Assess whether use of intraurethral 2% lidocaine jelly meaningfully impacts sensation during filling (especially, strong desire to void).
Time Frame: Within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
mL
  First Sensation | 17 [9 to 44] | 18 [11 to 37]
  First Urge to Void | 137 [86 to 191] | 107 [62 to 238]
  Strong Urge to Void | 243 [186 to 318] | 263 [161 to 396]
  Maximum Capacity | 344 [267 to 505] | 365 [275 to 450]

2. Secondary Outcome: Patient Perception of Pain/Discomfort as Indicated by Visual Analog Scale (Scale of 0-100 With 0 Being no Pain and 100 Being the Worst the Pain Imaginable).
Description: Determine whether the use of intraurethral lidocaine 2% jelly meaningfully impacts pain/discomfort measured by a visual analog scale during cystometry (catheter insertion and at maximum cystometric capacity), during pressure flow study (PFS), and post-procedure.
Time Frame: Change from cystometrogram 1 to cystometrogram 2 within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: mm on a VAS Pain Scale
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
mm on a VAS Pain Scale
  Catheter insertion | 7 [2 to 17.8] | 4.5 [1 to 20.2]
  Maximum capacity | 8 [4.2 to 25] | 10 [4 to 38]
  Pressure flow study | 7 [2 to 18] | 3 [0 to 8]
  Overall participant discomfort | 9 [2 to 21] | 4 [2 to 16]

3. Secondary Outcome: Provider Perception of Patient Pain/Discomfort as Indicated by Visual Analog Scale (Scale of 0-100 With 0 Being no Pain and 100 Being the Worst Pain Imaginable).
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts provider perception of patient discomfort.
Time Frame: Change from cystometrogram 1 to cystometrogram 2 within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: mm on a VAS Pain Scale
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
mm on a VAS Pain Scale | 9 [2 to 27] | 6 [2 to 16]

4. Secondary Outcome: Filling Metrics: Number of Participants With Detrusor Overactivity
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts the presence/absence of detrusor overactivity (bladder spasm) during urodynamic bladder testing. Detrusor overactivity was noted and compared between placebo and lidocaine jelly on UDS #2.
Time Frame: Cystometrogram 2 within same visit, approximately 90-120 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
Participants | 10 | 6

5. Secondary Outcome: Filling Metrics: Number of Participants With Normal Bladder Compliance
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts bladder compliance (change in volume/ change in detrusor pressure (Pdet)). Compliance in UDS #2 was noted and compared in both groups: water-based lubricant and intraurethral 2% lidocaine jelly. Results indicate how many participants in which normal compliance was observed. *There were 3 missing data values in our data.
Time Frame: Within same visit, approximately 90-120 minutes.
Population: *There were 3 missing data values in our data.
Measure: Count of Participants; unit: Participants
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 28 | 32
Participants | 28 | 32

6. Secondary Outcome: Voiding Metrics: Maximum Flow Rate
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts maximum flow rate (mL/sec).
Time Frame: Within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: mL/sec
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
mL/sec | 18.2 [11.6 to 25.4] | 16.5 [11.8 to 22.2]

7. Secondary Outcome: Voiding Metrics: Voiding Pattern (Normal vs. Intermittent/Interrupted vs Prolonged) as Perceived by Provider Interpretation of Pressure Flow Study During Voiding Based on Seconds to Void and Whether Urine Stream is Constant or Intermittent/Interrupted.
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts voiding pattern. Voiding pattern was assessed in UDS #2 and identified as either "normal", "prolonged", "intermittent", "interrupted" or a combination of those identifiers and compared between the two groups.
Time Frame: within same visit, approximately 90-120 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
Participants
  Normal | 3 | 3
  Intermittent | 15 | 21
  Interrupted | 14 | 18
  Prolonged | 17 | 24

8. Secondary Outcome: Voiding Metrics: Voided Volume and Post-void Residual
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts voided volume and post-void residual (mL) as recorded during UDS #2.
Time Frame: Within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
mL
  Voided Volume | 278 [174 to 400] | 318 [225 to 402]
  Post Void Residual | 29 [0 to 61] | 15 [0 to 66]

9. Secondary Outcome: Voiding Metrics: Percentage of Voiding Efficiency
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts voiding efficiency, which is calculated as the voided volume (mL) divided by the sum of the voided volume (mL) and the post-void residual volume (mL). Voiding efficiency was compared by treatment arm in UDS #2.
Time Frame: Cystometrogram 2 within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: percentage of voiding efficiency
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
percentage of voiding efficiency | 94.6 [72.2 to 100] | 95.9 [82.3 to 100]

10. Secondary Outcome: Voiding Metrics: Pdet Max
Description: Determine whether the use of intraurethral 2% lidocaine jelly meaningfully impacts Pdet Max (cm/H2O) on UDS #2.
Time Frame: Within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: cm/H2O
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
cm/H2O | 37 [26.5 to 46] | 28.5 [20 to 46.8]

11. Secondary Outcome: Voiding Metrics: Pdet Peak Flow
Description: Determine whether the use of intraurethral 2& lidocaine jelly meaningfully impacts Pdet Peak Flow (cm/H2O) on UDS #2.
Time Frame: Within same visit, approximately 90-120 minutes.
Measure: Median (Inter-Quartile Range); unit: cm/H2O
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
Number analyzed (Participants) | 30 | 33
cm/H2O | 20 [9 to 30] | 13 [7 to 18]

ADVERSE EVENTS:
Time Frame: Patients undergoing urodynamics were found to have positive urine cultures from sample sent immediately prior to the procedure. Patients were treated only if symptomatic. Treatment included antibiotic medication for 1 week.
Description: There were no deaths, all-cause mortality or serious adverse events. Other adverse events exceeding 5% frequency include asymptomatic bacteuria- presence of bacteria in urine without any urinary tract infection symptoms present.
Arm/Group | Water Based Lubricating Jelly | Lidocaine 2% Jelly
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 2/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Water Based Lubricating Jelly (N=30) | Lidocaine 2% Jelly (N=33)
asymptomatic bacteuria (Renal and urinary disorders) | 0 (0) | 2 (2) — Patient urine cultures came back positive for asymptomatic bacteuria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT04038099/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT04038099/ICF_001.pdf